CLINICAL TRIAL: NCT05301439
Title: Controlled Clinical Trial Of The Use Of Hall Technique In Deciduous Molars Affected By Extensive Caries Lesions. Follow Up Of 12 Months.
Brief Title: Use Of Hall Technique In Deciduous Molars Affected By Extensive Caries Lesions
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HallTechnique
Record Dates: First submitted 2022-03-16; First posted 2022-03-29 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Caries
MeSH Terms: interventions — Resins, Plant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical and radiographic evaluations of the complete removal of the carious lesion will be performed by two calibrated examiners blinded to the allocation of teeth to the different groups. Also, calibrated examiners, who will not be performing the restorations and therefore will be blind to the groups, will perform the assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Restoration Group (Experimental): Participants in this group will receive the universal adhesive restorative procedure combined with condensable bulk fill resin, for the restoration of the cavited teeth.
  Interventions: Procedure: Restoration with Resin
- Hall Technique Group (Experimental): Participants in this group will receive the Hall Technique with steel crowns for the restoration of the cavited teeth.
  Interventions: Procedure: Hall Technique
- Steel Crown with Conventional Technique Group (Experimental): Participants in this group will receive steel crowns with conventional technique for the restoration of the cavited teeth.
  Interventions: Procedure: Conventional Steel Crown

INTERVENTIONS:
Procedure: Restoration with Resin — Prophylaxis with prophylactic paste and rubber cup. Relative isolation (lip retractor, cotton roll and saliva sucker). Selective removal of carious tissue with dentin spoons at the dentin-enamel junction.
  Cleaning the cavity with water. Application of the Universal Adhesive System (Shofu). Excess removal. Application of a new layer of adhesive system. Light rubbing and excess removal. Photoactivation - 20s. Insert Bulk Fill Resin (Shofu) in 4mm increments. Photoactivation for 20". Preservation. Clinical and radiographic control at 1, 3, 6 and 12 months.
  Arms: Restoration Group
Procedure: Hall Technique — Prophylaxis with prophylactic paste and rubber cup. Relative isolation (lip retractor, cotton roll and saliva sucker). Clinical evaluation through inspection of the texture of the remaining dentin with a rounded exploratory probe.
  Cleaning the cavity with water. Take drying. Proof of the steel crown. Relative isolation. Filling the inner part of the crown with bioactive resin cement or glass ionomer cement for cementation.
  Clinical and radiographic control at 1, 3, 6 and 12 months.
  Arms: Hall Technique Group
Procedure: Conventional Steel Crown — * Prophylaxis;
  * Relative isolation;
  * The preparation of the tooth will be performed conventionally with reduction of the occlusal, mesial and distal surface of 1 to 1.5 mm and selective removal of the decayed tissue;
  * Cleaning the cavity with water;
  * Slight drying;
  * Trial of steel crown;
  * Relative isolation;
  * Filling the inner part of the crown with bioactive resin cement or glass ionomer cement for cementation.
  * Clinical and radiographic control at 1, 3, 6 and 12 months.
  Arms: Steel Crown with Conventional Technique Group

SUMMARY:
Despite preventive treatments and the promotion of oral health, dental caries is one of the most prevalent chronic diseases in the population and treatment of caries lesions in deciduous teeth is a fundamental procedure aimed at increasing the resistance of the remaining tooth structure to preserve the permanent dentition. The present study aims to make a clinical evaluation of the Hall Technique compared to direct restorations with universal adhesives and bulk fill resins in large destruction of deciduous teeth. 90 children between 5 and 10 years old, healthy, of both sexes, without distinction of race, enrolled in the clinics of Universidade Metropolitana de Santos-UNIMES will be selected. The in-office treatments will be carried out by a trained researcher, according to the manufacturer's instructions for each material and scientific evidence on the respective topic. Participants will be divided into 03 groups according to the proposed treatments. Group 1 - Universal adhesive restorative procedure + condensable bulk fill resin; Group 2 - Hall Technique with Shofu steel crowns and Group 3 - Steel crown with conventional technique. The evaluated outcomes will be: effectiveness of the technique and longevity of the restorations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy child, without systemic changes;
2. Good behavior;
3. Clinically, present at least two deciduous molars with caries in dentin involving more than three surfaces, with vision and direct access, without signs and symptoms of pulp involvement.

Exclusion Criteria:

1. Children with any serious systemic disorder;
2. Lack of cooperation.
3. Clinically present at least one deciduous molar with carious lesion in the dentin involving signs and symptoms of pulpal involvement.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Changes in the Longevity Of Restorations | Three, 6 and 12 months after treatment.
  Steel restorations and crowns will be classified according to the criteria in the following scores: FDI criterion (clinically very good, clinically good, clinically sufficient/satisfactory, clinically unsatisfactory, clinically poor).

SECONDARY OUTCOMES:
Changes in the biofilm index | Baseline, 3, 6, and 12 months after treatment.
  The presence of biofilm will be evaluated through the Simplified Oral Hygiene Index (OHI-S).
Changes in Salivary PH | Baseline, 6, and 12 months after treatment.
  Participants will be asked to spit into a collection pot, in which the pH will be measured with measuring stripes.
Changes in The Presence of Caries Lesions | Baseline, 6, and 12 months after treatment.
  A clinical evaluation in the search of carious lesions will be performed.
Technique Perfomance Time Duration | During the procedure.
  To take the time, a previously calibrated digital stopwatch will be used.